CLINICAL TRIAL: NCT04445181
Title: Canadian REgistry of Chronic Kidney Disease in Diabetes Outcomes (CREDO) Study
Brief Title: A Study Using the LMC Diabetes Registry to Learn More About Chronic Kidney Disease (CKD) in Canadian Patients With Type 2 Diabetes (T2D)
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21190
Record Dates: First submitted 2020-06-21; First posted 2020-06-24 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Chronic Kidney Disease in Type 2 Diabetes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with T2D: Active patients (defined as patients seen by an LMC endocrinologist between January 1, 2019 and December 31, 2019) with T2D (Type 2 Diabetes). Among the patients with T2D, those identified with CKD will be included in the renal registry.
  Interventions: Drug: The physician's prescription in routine clinical practice
- Healthcare providers: Healthcare providers caring for patients with CKD and T2D.

INTERVENTIONS:
Drug: The physician's prescription in routine clinical practice — This is an Observational study that will not involve prescription of the drugs.
  Groups: Patients with T2D

SUMMARY:
In people with type 2 diabetes (T2D), the body does not make enough of a hormone called insulin or does not use insulin well. This results in high blood sugar levels.

People with T2D are at a higher risk of having a condition called chronic kidney disease (CKD). In people with CKD, the kidneys become damaged and do not work as they should. People with CKD can have trouble breathing and often have swelling in their arms and legs, and high blood pressure.

People who have CKD and T2D are more likely to have other medical problems, such as heart disease.

There are many treatments available to patients who have CKD and T2D. But, researchers need more information about how doctors in Canada are deciding which treatment to give these patients.

In this study, the researchers will review health information from men and women with T2D who visited a doctor in 2019 and had check-ups for at least 6 months. The health information will be taken from a Canadian registry (or database) owned by LMC Diabetes & Endocrinology. The registry contains information from people that went to an LMC clinic. In this study, the researchers will learn how many of these people had T2D and CKD. They will learn the treatments these people received, and if they had other related medical problems. The researchers will also use surveys to ask the doctors about why they chose certain treatments.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of T2D as captured in the LMC EMR system
* Assessed by an LMC endocrinologist between January 1, 2019 and December 31, 2019
* Followed by an LMC endocrinologist for ≥ 6 months prior to inclusion in the cohort
* Informed consent to use patient medical record data for research purposes was provided

Among patients who meet the inclusion criteria, estimated glomerular filtration rate (eGFR) ≤ 60 ml/min/1.73 m^2 and/or urine albumin-to-creatinine ratio (uACR) ≥ 2 mg/mmol will be used to identify the cohort of patients with T2D and CKD

Exclusion Criteria:

- Any patients with documented non-diabetic etiology for renal disease will be excluded from the numerator (number of patients with CKD and T2D) when determining the primary endpoint

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include active LMC patients with T2D. This population will be used to determine the prevalence of CKD in patients with T2D. Patients identified with T2D and CKD will form the cohort for all subsequent analysis.
Sampling Method: Non-Probability Sample
Enrollment: 14873 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with CKD in a large T2D population | Retrospectively analysis between January 1, 2019 and December 31, 2019
  The data will be retrieved from the LMC Diabetes Registry, a Pan-Canadian registry of diabetes community-based specialist practices and used to develop a renal registry to investigate the primary objectives of the study

SECONDARY OUTCOMES:
Proportion of patients using the different therapies | Retrospectively analysis between January 1, 2019 and December 31, 2019
  The therapies are: ACEi, ARBs, ACEi/ARBs, MRAs, GLP-1 RA and SGLT2i
Proportion of patients with stage 1 CKD with moderate or greater albuminuria, stage 2 CKD with moderate or greater albuminuria, stage 3a CKD, stage 3b CKD, stage 4 CKD and stage 5 CKD in accordance with Canadian clinical practice guidelines | Retrospectively analysis between January 1, 2019 and December 31, 2019
  Stage 1 CKD: eGFR (estimated glomerular filtration rate) ≥ 90 ml/min/1.73 m^2 Stage 2 CKD: eGFR between 60-89 ml/min/1.73 m^2 Stage 3a CKD: eGFR between 45-59 ml/min/1.73 m^2 Stage 3b CKD: eGFR between 30-44 ml/min/1.73 m^2 Stage 4 CKD: eGFR between 15-29 ml/min/1.73 m^2 Stage 5 CKD: eGFR <15 ml/min/1.73 m^2
Proportion of patients with microalbuminuria and macroalbuminuria, in accordance with Canadian clinical practice guidelines | Retrospectively analysis between January 1, 2019 and December 31, 2019
  Microalbuminuria: uACR (urine albumin-to-creatinine ratio) 2-20 mg/mmol Macroalbuminuria: uACR > 20 mg/mmol
Proportion of patients within each albuminuria category (A1, A2 or A3), in accordance with KDIGO clinical practice guidelines | Retrospectively analysis between January 1, 2019 and December 31, 2019
  KDIGO = Kidney Disease: Improving Global Outcomes
Laboratory values for patients using either no therapy or using a therapy for ≥ 6 months | Retrospectively analysis between January 1, 2019 and December 31, 2019
  Laboratory values including glucose, glycated hemoglobin (HbA1c), lipids, creatinine, electrolytes, eGFR, and uACR
Proportion of patients with different comorbidities | Retrospectively analysis between January 1, 2019 and December 31, 2019
  Comorbidities like hypertension, dyslipidemia, microvascular disease, macrovascular disease
Proportion of healthcare provider prescriptions of RAS therapies (ACEi/ARB) used to treat hypertension, heart failure, coronary artery disease, CKD, or other condition | On the day of healthcare provider completes a questionnaire
  RAS: renin angiotensin system ACEi: angiotensin converting enzyme inhibitors ARB: angiotensin receptor blocker
  Healthcare providers will complete a questionnaire to determine their rationale for use of common therapies for CKD in T2D
Proportion of healthcare provider prescriptions of GLP-1 RA used to treat glycemia management, hypertension, heart failure, coronary artery disease, CKD or other condition | On the day of healthcare provider completes a questionnaire
  GLP-1 RA: glucagon-like peptide-1 receptor agonist
  Healthcare providers will complete a questionnaire to determine their rationale for use of common therapies for CKD in T2D
Proportion of healthcare provider prescriptions of MRAs used to treat hypertension, heart failure, coronary artery disease, CKD or other condition | On the day of healthcare provider completes a questionnaire
  MRAs: mineralocorticoid receptor antagonists
  Healthcare providers will complete a questionnaire to determine their rationale for use of common therapies for CKD in T2D
Proportion of healthcare provider prescriptions of SGLT2i used to treat glycemia management, hypertension, heart failure, coronary artery disease, CKD or other condition | On the day of healthcare provider completes a questionnaire
  SGLT2i: sodium-glucose co-transporter-2 inhibitors
  Healthcare providers will complete a questionnaire to determine their rationale for use of common therapies for CKD in T2D

CONTACTS AND LOCATIONS:
Locations (1):
- A Database, A Database, Canada

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Chu L, Fuller M, Jervis K, Ciaccia A, Abitbol A. Prevalence of Chronic Kidney Disease in Type 2 Diabetes: The Canadian REgistry of Chronic Kidney Disease in Diabetes Outcomes (CREDO) Study. Clin Ther. 2021 Sep;43(9):1558-1573. doi: 10.1016/j.clinthera.2021.07.015. Epub 2021 Aug 21. PMID 34426012
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/